CLINICAL TRIAL: NCT01356875
Title: Phase II Clinical Trial for Treatment of Myelodysplastic Syndromes Comparing Hydralazine / Ac.Valproico and Supportive Care in Patients Not Candidates, Refractory and / or Intolerant to Intensive Chemotherapy
Brief Title: Treatment of Myelodysplastic Syndromes Comparing Hydralazine/Ac. Valproic and Supportive Care in Patients Not Candidates, Refractory and/or Intolerant to Intensive Chemotherapy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Basque Health Service (Other Government)
Responsible Party: Breno Moreno De Gusmao, Osakidetza/Basque Health Service
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SMD-TXAGO
Record Dates: First submitted 2011-05-18; First posted 2011-05-20 (Estimated); Last update posted 2011-05-20 (Estimated); Status verified 2011-04

CONDITIONS: Myelodysplastic Syndrome
Keywords: myelodysplastic syndrome; Transfusion; Hydralazine; valproic acid
MeSH Terms: conditions — Myelodysplastic Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- HIDRA/VPA (Experimental): In each cycle (30 days), Hydralazine 50mg tablets every 12 hours and Valproic 500mg tablets every 8 hours will be administrated orally to HYDRA / VPA group.Each patient will receive 6 cycles of hydralazine and valproic acid.
  Interventions: Drug: HIDRA/VPA
- best supportive care (BSC) (Active Comparator): The support group will be receive transfusional BSC, erythropoietin and / or G-CSF as determined by the physician.
  Interventions: Drug: BSC

INTERVENTIONS:
Drug: BSC — The support group will be receive transfusional BSC, erythropoietin and / or G-CSF as determined by the physician.
  Arms: best supportive care (BSC)
Drug: HIDRA/VPA — In each cycle (30 days), Hydralazine 50mg tablets every 12 hours and Valproic 500mg tablets every 8 hours will be administrated orally to HYDRA / VPA group.Each patient will receive 6 cycle.
  Arms: HIDRA/VPA

SUMMARY:
Transfusional dependence has been associated closely and independently with low survival in patients with myelodysplastic syndrome (MDS), especially in patients at low risk according to IPSS. Treatment of patients with hydralazine + valproic acid as an alternative to treatment with 5-azacytidine has lower cost and possibly as effective with fewer side effects. The objective of this phase II study is to determine the effectiveness of combination therapy with hydralazine + Ac. Valproic compared with best supportive care. The investigators will select 42 patients per group, and after 14 weeks of treatment the investigators will study in both groups the hematological response (transfusion-dependent, hemoglobin, cytogenetics and morphology) and treatment safety (adverse reactions and vital signs) to 1 year after starting treatment. The concentration of hemoglobin, the number of transfusions, platelets, neutrophils and other continuous variables in both groups will be compared by Student t or Mann-Whitney, as appropriate. For comparison of cytogenetic and morphological response and other categorical variables between groups Chi square will be used. And within each group the investigators will compare each of these variables before and after treatment by t-test for paired data or Wilcoxon test.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to understand and voluntarily sign the consent form.
2. Age ≥ 18 years at the time of signing the informed consent form.
3. Ability and willingness to meet the schedule of study visits and other protocol requirements.
4. Documented diagnosis of SMDs according to the criteria of disease risk IPSS intermediate-2, high risk or any risk with transfusion requirements.
5. Transfusion-dependent anemia erythrocytes defined as the absence of a period of 56 consecutive days without transfusion of red blood cells for at least 112 days prior (16 weeks).
6. Engage both women and men to use highly effective contraception.
7. Patients are not candidates for treatment with azacitidine or chemotherapy

Exclusion Criteria:

* Patients who have any of these exclusion criteria may not be included in the trial:

  1. Pregnant or breastfeeding.
  2. After hematopoietic stem cell transplantation.
  3. Patients with vitamin B12 deficiency, Folic Acid and Iron
  4. Any severe psychiatric illness or condition that prevents the patient sign the consent form for the patient or involves an unacceptable risk in case of participating in the study.
  5. Hypersensitivity to hydralazine and / or AC. Valproic

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2011-09; Primary Completion 2014-09 (Estimated); Study Completion 2015-01 (Estimated)

PRIMARY OUTCOMES:
change in hemoglobin from baseline in patients who express an erythroid response. | 8 weeks
  Independence RBC transfusion requirement for ≥ 8 weeks (56 days) followed by treatment at any time.

SECONDARY OUTCOMES:
Erythroid response according to the criteria of the international working group of SMDs at 24 weeks | 24 weeks
  Number and type of administered blood transfusions, time between the last transfusion prior to inclusion in the study and the first transfusion after the 8 weeks of treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Txagorritxu Hospital, Vitoria-Gasteiz, Alava, Spain